CLINICAL TRIAL: NCT03904823
Title: An Open, Single-arm, Multi-center, Phase 2 Clinical Trial of Famitinib Combined With Epidermal Growth Factor Receptor (EGFR) Inhibitor HS-10296 in Patients With Advanced EGFR-mutant Non-Small Cell Lung Cancer (NSCLC)
Brief Title: A Study of Famitinib in Combination With HS-10296 in Patients With EGFR-mutant NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMTN-II-203-NSCLC
Record Dates: First submitted 2019-04-02; First posted 2019-04-05 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-06

CONDITIONS: EGFR-mutant Non-Small Cell Lung Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- famitinib, HS-10296 (Experimental)
  Interventions: Drug: famitinib po; Drug: HS-10296 po

INTERVENTIONS:
Drug: famitinib po — Patients would be treated with famitinib po combined with HS-10296 po till progression disease or withdrawal from the study.
Drug: HS-10296 po — Patients would be treated with famitinib po combined with HS-10296 po till progression disease or withdrawal from the study.

SUMMARY:
The study is being conducted to evaluate the efficacy, safety and tolerability of famitinib combined with HS-10296 in subjects with advanced EGFR-mutant NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Subject's written informed consent obtained prior to any process, sampling, or analysis related to the study.
* Male or female, no less than 18 years old.
* Confirmed as NSCLC by histology or cytology.
* Locally advanced or metastatic NSCLC and not suitable for radical surgery or radiotherapy.
* Have not received EGFR Tyrosine Kinase Inhibitor (TKI) therapy.
* At least one baseline tumor lesion.
* Can swallow pills normally.
* Eastern Cooperative Oncology Group (ECOG) performance status 0~1 points, expected survival≥12 weeks.
* Adequate organ function.

Exclusion Criteria:

* Clinically symptomatic central nervous system metastases.
* Ascites, pleural effusion or pericardial effusion with clinical symptoms.
* Other malignant tumors in the past 5 years or at the same time.
* High blood pressure which are not well controlled.
* Heart disease that are not well controlled.
* Coagulation dysfunction, bleeding tendency or receiving thrombolysis or anticoagulant therapy.
* History of bleeding.
* Known hereditary or acquired bleeding and thrombophilia.
* Any serious or uncontrolled ocular lesion.
* Interstitial lung disease or non-infectious pneumonia treated with corticosteroids.
* Congenital or acquired immunodeficiency.
* Other factors that may affect the results of the study or cause the study to be terminated midway.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2019-04-25 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | From the start of treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Based on response evaluation criteria in solid tumors 1.1 (RECIST 1.1)

SECONDARY OUTCOMES:
Depth of Response (DepOR) | From the start of treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Percentage of total target lesion diameter reduced from baseline when at best overall response
Duration of Response (DOR) | From the first partial response or complete response until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Based on response evaluation criteria in solid tumors 1.1 (RECIST 1.1)
Disease Control Rate (DCR) | From the start of treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Based on response evaluation criteria in solid tumors 1.1 (RECIST 1.1)
Clinical Benefit Ratio (CBR) | From the start of treatment to 6 months
  Based on response evaluation criteria in solid tumors 1.1 (RECIST 1.1)
12-month-PFS | From the start of treatment to 12 months
  12-month-progression free survival rate
Progression-Free-Survival (PFS) | up to 2 years
  Based on response evaluation criteria in solid tumors 1.1 (RECIST 1.1)
Number of Participants with Clinically significant toxicity | First cycle (21 days)
  Number of Participants with Clinically significant toxicity per National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0
Rate of Adverse Events and Serious Adverse Events | From the first drug administration to within 30 days after the last dose
  Rate of Adverse Events and Serious Adverse Events per National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Caicun Zhou, PhD, Principal Investigator — Shanghai Pulmonary Hospital, Shanghai, China
Locations (1):
- Tongji University, Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China